CLINICAL TRIAL: NCT04928131
Title: Opioid Use Among Patients With Pain Syndromes Commonly Seeking Surgical Consultation
Brief Title: Risk Factors for Long-term Opioid Use
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cindy Kin, Assistant Professor of Surgery, Stanford University
Other Study IDs: 43803
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pain Syndrome
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anorectal: Patients presenting with anorectal pain.
  Interventions: Other: No intervention - retrospective observational cohort study
- TMJ: Patients presenting with temporomandibular joint pain.
  Interventions: Other: No intervention - retrospective observational cohort study
- Foot/Ankle: Patients presenting with foot and ankle pain.
  Interventions: Other: No intervention - retrospective observational cohort study

INTERVENTIONS:
Other: No intervention - retrospective observational cohort study

SUMMARY:
Surgeons often see patients with pain to exclude organic pathology and consider surgical treatment. We examined factors associated with long-term opioid therapy among patients with foot/ankle, anorectal, and temporomandibular joint pain to aid clinical decision making.

Using the IBM MarketScan® Research Database, we conducted a retrospective cohort analysis of patients aged 18-64 with a clinical encounter for foot/ankle, anorectal, or temporomandibular joint pain (January 2007-September 2015). Multivariable logistic regression was used to estimate adjusted odds ratios for factors associated with long-term opioid therapy, including age, sex, geographic region, pain condition, psychiatric diagnoses, and surgical procedures in the previous year.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* at least one encounter for anorectal, foot/ankle, or TMJ pain
* Marketscan continuous enrollment for 1 year prior and 1 year after the index pain encounter

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: adult patients enrolled in private health insurance included within the Marketscan database, who generated at least one insurance claim for anorectal, foot/ankle, or TMJ pain.
Sampling Method: Non-Probability Sample
Enrollment: 1500392 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Long-term opioid use | >90 days of opioid supply
  opioid prescriptions for 3 months.

SECONDARY OUTCOMES:
new long-term opioid use | >90 days of opioid supply
  Opioid prescriptions for over 3 months in patients who have not had prior opioid prescriptions.